CLINICAL TRIAL: NCT00087139
Title: Phase II Study of a Weekly Schedule of BMS-247550 for Patients With Hormone Refractory Prostate Cancer
Brief Title: Ixabepilone in Treating Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00548; NCI-2009-00548 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000372946; E3803; E3803 (Other: Eastern Cooperative Oncology Group); E3803 (Other: CTEP); U10CA021115 (NIH)
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Results first posted 2012-12-27 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2013-04

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — ixabepilone

ARMS (1):
- Arm I (Experimental): Patients are stratified according to prior chemotherapy (none vs 1 prior taxane-containing regimen vs 2 prior cytotoxic regimens).
  Patients receive ixabepilone IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: ixabepilone

INTERVENTIONS:
Drug: ixabepilone — Given IV
  Other Names: BMS-247550; epothilone B lactam; Ixempra

SUMMARY:
Drugs used in chemotherapy, such as ixabepilone, work in different ways to stop tumor cells from dividing so they stop growing or die. This phase II trial is studying how well ixabepilone works in treating patients with metastatic prostate cancer that has not responded to previous hormone therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the effect on percent with a 50% decrease in PSA response in patients with metastatic prostate cancer who have progressed on androgen ablation therapy and are classified into 1 of 3 separate categories:

1. Never received prior chemotherapy/cytotoxic therapy
2. Received prior taxane-based regimen
3. Received 2 prior cytotoxic chemotherapy regimens (including, but not limited to, prior taxane and anthracyclines)

SECONDARY OBJECTIVES:

I. Determine measurable disease response in patients with measurable disease treated with this drug and overall response rate.

II. Determine the toxic effects of this drug in these patients. III. Determine the duration of PSA and measurable disease response in patients treated with this drug.

IV. Determine the expression of p53, multidrug resistance protein, and Bcl-2 by immunohistochemistry in the primary tumors of patients treated with this drug.

OUTLINE: This is a multicenter study. Patients are stratified according to prior chemotherapy (none vs 1 prior taxane-containing regimen vs 2 prior cytotoxic regimens).

Patients receive ixabepilone IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Metastatic disease
* Evidence of disease progression (e.g., new lesions on bone scan or new/enlarging lesions on CT scan) OR rising prostate-specific antigen (PSA) within the past 4 weeks
* Radiologic evidence of hydronephrosis alone is not considered evidence of metastatic disease (e.g., increasing PSA)
* Patients with bone metastases only (i.e., lacking soft tissue disease) must have a PSA level >= 10 ng/mL within the past week
* Patients with stable disease and rising PSA must show 2 consecutive rises in PSA measurements taken at least 2 weeks apart
* Most recent PSA level must be obtained within the past 4 weeks
* Disease progression after prior anti-androgen withdrawal must be confirmed by a rising PSA after the 4-6 week washout period (e.g., PSA level higher than the last PSA obtained while on anti-androgen therapy)
* Failed prior bilateral orchiectomy or other primary hormonal therapy
* Patients who have not undergone bilateral orchiectomy must continue on luteinizing hormone-releasing hormone (LHRH) agonist therapy (e.g., leuprolide or goserelin) or LHRH antagonist (e.g., abarelix) during study treatment AND must have a serum testosterone level =< 50 ng/dL within the past 4 weeks to confirm androgen suppression
* ECOG 0-2
* Granulocyte count >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* WBC >= 4,000/mm^3
* SGPT =< 2 times upper limit of normal
* Bilirubin =< 1.5 mg/dL
* INR normal
* Creatinine =< 1.5 mg/dL
* Creatinine clearance >= 50 mL/min
* No New York Heart Association class III-IV heart disease
* No myocardial infarction within the past 6 months
* No active angina pectoris
* No evidence of ventricular dysrhythmias or other unstable arrhythmia
* Rate-controlled atrial fibrillation allowed provided the patient is asymptomatic
* No other malignancy within the past 5 years except curatively treated nonmelanoma skin cancer
* No serious medical illness or active infection that would preclude study participation
* No concurrent prophylactic filgrastim (G-CSF)
* No more than 2 prior cytotoxic chemotherapy regimens for hormone-refractory disease
* At least 4 weeks since prior chemotherapy with a taxane-based regimen, mixantrone, or another cytotoxic chemotherapy regimen provided there is evidence of progressive disease
* At least 4 weeks since prior flutamide AND continued evidence of progressive disease
* At least 6 weeks since prior bicalutamide or nilutamide AND continued evidence of progressive disease
* At least 4 weeks since prior estrogen or estrogen-like agents (e.g., PC-SPES, saw palmetto, or other herbal products which may contain phytoestrogens)
* At least 4 weeks since prior hormonal therapy, including megestrol, finasteride, ketoconazole, or systemic corticosteroids
* No concurrent estrogen or estrogen-like agents (e.g., PC-SPES, saw palmetto, or other herbal products which may contain phytoestrogens)
* More than 4 weeks since prior radiotherapy
* No prior strontium chloride Sr 89 or samarium Sm 153 lexidronam pentasodium
* No other prior radioisotope
* No concurrent radiotherapy for pain control
* No more than 1 prior experimental (non-cytotoxic) therapy AND evidence of progressive disease
* At least 4 weeks since prior experimental therapy
* Concurrent bisphosphonates (e.g., pamidronate or zoledronate) allowed provided treatment was initiated at least 4 weeks ago and there is evidence of progressive disease
* No other concurrent investigational agents
* No concurrent therapeutic warfarin
* Concurrent prophylactic or therapeutic doses of low molecular weight heparin allowed provided criterion for INR is met
* No carcinomatous meningitis or brain metastases
* Fertile patients must use effective contraception
* No peripheral neuropathy > grade 1

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2004-09; Primary Completion 2009-04 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Liu, Principal Investigator — Eastern Cooperative Oncology Group
Locations (162):
- United States (162):
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Saint Francis Hospital - Wilmington, Wilmington, Delaware
  - Edna Williams Cancer Center at the Baptist Cancer Institute, Jacksonville, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Alexian Brothers Medical and Cancer Center, Elk Grove Village, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Vigliotti, Antonio, P.G. M.D. (UIA Investigator), Moline, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Clinic-Urbana Main, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - Indiana University Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center - Mishawaka, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Association, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Community Memorial Hospital, Missouri Valley, Iowa
  - Burgess Memorial Hospital, Onawa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Eastern Cooperative Oncology Group, Boston, Massachusetts
  - Morton Hospital and Medical Center, Taunton, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium Community Clinical Oncology Program, Ann Arbor, Michigan
  - Oakwood Hospital, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Essentia Health Duluth Clinic CCOP, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Fremont Area Medical Center, Fremont, Nebraska
  - Bryan LGH Medical Center West, Lincoln, Nebraska
  - Bryan LGH Medical Center East, Lincoln, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Ocean Medical Center, Brick, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - Cancer Institute of New Jersey At Hamilton, Hamilton, New Jersey
  - Mountainside Hospital, Montclair, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital of Burlington County, Mount Holly, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Virtua West Jersey Hospital Voorhees, Voorhees Township, New Jersey
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Montefiore Medical Center-Wakefield Campus, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Mercy Medical Center, Canton, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - Mainline Health CCOP, Wynnewood, Pennsylvania
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran, La Crosse, Wisconsin
  - UW Health Oncology - 1 South Park, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on September 16, 2004 and terminated on February 4, 2009 after reaching its accrual goal. A total of 124 patients were recruited from ECOG member institutions.
Groups:
- Ixabepilone - no Prior Chemo; Ixabepilone - Prior Taxane; Ixabepilone - Two Prior Chemo: All patients on this study received the same treatment but were categorized into 3 strata, including the no prior chemo stratum, the prior taxane stratum, and two prior chemo stratum. Only eligible and treated patients are included in the analysis.
Period: Overall Study
Arm/Group | Ixabepilone - no Prior Chemo | Ixabepilone - Prior Taxane | Ixabepilone - Two Prior Chemo
Started | 39 | 49 | 36
Treated | 39 | 48 | 36
Eligible and Treated | 35 | 42 | 32
Patients for the Analysis of PSA Respons | 30 | 34 | 22
Patients With Measurable Disease | 22 | 25 | 24
Patients With PSA Response | 10 | 8 | 4
Patients w/ Measurable Disease Response | 5 | 2 | 0
Completed | 0 | 0 | 0
Not Completed | 39 | 49 | 36
Not completed — Adverse Event | 18 | 17 | 13
Not completed — Death | 2 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 2
Not completed — Physician Decision | 1 | 1 | 1
Not completed — Disease progression | 9 | 19 | 12
Not completed — Ineligible | 4 | 7 | 4
Not completed — Symptomatic deterioration | 1 | 1 | 3
Not completed — Use of coumadin | 1 | 0 | 0
Not completed — Response achieved | 0 | 1 | 0
Not completed — Extradural disease | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ixabepilone - no Prior Chemo | Ixabepilone - Prior Taxane | Ixabepilone - Two Prior Chemo | Total
Number analyzed (Participants) | 35 | 42 | 32 | 109
Age, Continuous [Median (Full Range); unit: years] | 72 [45 to 82] | 69 [50 to 81] | 67.5 [49 to 90] | 70 [45 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 35 | 42 | 32 | 109

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With PSA Response
Description: PSA response is defined as a decline from baseline value by >=50%, or normalization of PSA (PSA < 0.2 ng/lm), confirmed by a second measurement >= 4 weeks later. The proportion of patients with PSA response was reported separately for 3 strata. Additional patients accrued to this study were not included in this analysis.
Time Frame: Every 4 weeks during treatment; then every 3 months if <2 years from study entry; then every 6 months if 2-5 years from study entry
Population: If the regimen demonstrated a PSA response rate specified in the protocol, additional patients would be entered so the total number of eligible patients with measurable disease in each stratum is 25. But the PSA response rate was only calculated among the first cohort of patients, not including the additional patients with measurable disease.
Measure: Number (90% Confidence Interval); unit: Proportion of participants
Arm/Group | Ixabepilone - no Prior Chemo | Ixabepilone - Prior Taxane | Ixabepilone - Two Prior Chemo
Number analyzed (Participants) | 30 | 34 | 22
Proportion of participants | 0.33 [0.19 to 0.5] | 0.24 [0.12 to 0.38] | 0.18 [0.06 to 0.37]

2. Secondary Outcome: Proportion of Patients With Measurable Disease Response (Best Overall Response)
Description: Only patients with measurable disease were included in this analysis. The proportion of patients with measurable disease response (based on RECIST: Response Evaluation Criteria in Solid Tumors) was reported separately for 3 strata.
  Per RECIST criteria, Complete response (CR)= disappearance of all target and nontarget lesions Partial response (PR)= >=30% decrease in the sum of the longest diameters of target lesions from baseline, and persistence of one or more non-target lesion(s) and/or the maintenance of tumor marker level above the normal limits.
  Objective response = CR + PR
Time Frame: Every 8 weeks during treatment; then every 3 months if <2 years from study entry; then every 6 months if 2-5 years from study entry
Population: Only patients with measurable disease were included in this analysis.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Ixabepilone - no Prior Chemo | Ixabepilone - Prior Taxane | Ixabepilone - Two Prior Chemo
Number analyzed (Participants) | 22 | 25 | 24
proportion of participants | 0.23 [0.09 to 0.42] | 0.08 [0.01 to 0.23] | 0 [0.0 to 0.12]

3. Secondary Outcome: Duration of PSA Response
Description: Duration of PSA response was defined as the time from the date of onset of PSA response until the date the criteria were met for PSA progression. Only patients with a PSA response were included in this analysis. The results were reported separately for 3 strata.
Time Frame: as for outcome 1
Population: If the regimen demonstrated a PSA response rate specified in the protocol, additional patients would be entered so the total number of eligible patients with measurable disease in each stratum is 25. But the PSA response related analysis was only done among the first cohort of patients, not including the additional patients with measurable disease.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ixabepilone - no Prior Chemo | Ixabepilone - Prior Taxane | Ixabepilone - Two Prior Chemo
Number analyzed (Participants) | 10 | 8 | 4
Months | 6.0 [1.8 to 8.0] | 7.6 [4.1 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for the assessment. | NA [NA to NA] — The median and 95% confidence interval were not calculable because none of them had progression at the final time point for the assessment.

4. Secondary Outcome: Duration of Measurable Disease Response
Description: Duration of measurable disease response was defined as the time from the date when measurement criteria were met for complete or partial response, whichever status was recorded first, until the first date that recurrent or progressive disease was objectively documented based on RECIST (Response Evaluation Criteria in Solid Tumors). Only patients with measurable disease response were included in this analysis.
Time Frame: as for outcome 2
Population: Only patients with measurable disease response were included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ixabepilone - no Prior Chemo | Ixabepilone - Prior Taxane | Ixabepilone - Two Prior Chemo
Number analyzed (Participants) | 5 | 2 | 0
Months | 5.1 [3.0 to 9.4] | 3.7 [NA to NA] — The lower and upper limits of the 95% confidence interval were not calculable because an insufficient number of participants reached the event at the final time point for the assessment. |

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment.
Groups:
- Ixabepilone: All patients who received protocol therapy, regardless of eligibility, were evaluated for toxicities.
Arm/Group | Ixabepilone
Serious Adverse Events (participants affected / at risk) | 90/123
Other Adverse Events (participants affected / at risk) | 122/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone (N=123)
Allergic reaction (Immune system disorders) | 1
Hearing: patients without baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 1
Anemia (Blood and lymphatic system disorders) | 8
Leukopenia (Investigations) | 27
Lymphopenia (Investigations) | 4
Neutropenia (Investigations) | 22
Thrombocytopenia (Investigations) | 1
Supraventricular arrhythmia NOS (Cardiac disorders) | 1
PVCs (Cardiac disorders) | 1
Hypotension (Vascular disorders) | 1
Fatigue (General disorders) | 28
Anorexia (Metabolism and nutrition disorders) | 12
Constipation (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 6
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 7
Ileus (Gastrointestinal disorders) | 2
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 3
Infection w/ Gr0-2 neutropenia, catheter (Infections and infestations) | 1
Infection w/ Gr0-2 neutropenia, lung (Infections and infestations) | 3
Infection w/ Gr0-2 neutropenia, skin (Infections and infestations) | 1
Duodenum, hemorrhage (Gastrointestinal disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 2
Ataxia (Nervous system disorders) | 4
CNS cerebrovascular ischemia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Neuropathy-motor (Nervous system disorders) | 13
Neuropathy-sensory (Nervous system disorders) | 32
Syncope (Nervous system disorders) | 4
Bone, pain (Musculoskeletal and connective tissue disorders) | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 3
Joint, pain (Musculoskeletal and connective tissue disorders) | 1
Neuropathic, pain (Nervous system disorders) | 2
Pain NOS (General disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone (N=123)
Anemia (Blood and lymphatic system disorders) | 112
Leukopenia (Investigations) | 84
Neutropenia (Investigations) | 51
Thrombocytopenia (Investigations) | 27
Hypotension (Vascular disorders) | 11
Fatigue (General disorders) | 89
Insomnia (Psychiatric disorders) | 21
Weight loss (Investigations) | 17
Alopecia (Skin and subcutaneous tissue disorders) | 45
Nail changes (Skin and subcutaneous tissue disorders) | 14
Rash/desquamation (Skin and subcutaneous tissue disorders) | 11
Anorexia (Metabolism and nutrition disorders) | 56
Constipation (Gastrointestinal disorders) | 29
Dehydration (Metabolism and nutrition disorders) | 10
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 41
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 15
Nausea (Gastrointestinal disorders) | 56
Taste disturbance (Nervous system disorders) | 31
Vomiting (Gastrointestinal disorders) | 30
Edema: limb (General disorders) | 15
ALT increased (Investigations) | 11
AST increased (Investigations) | 30
Bilirubin increased (Investigations) | 11
Creatinine increased (Investigations) | 18
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 11
Dizziness (Nervous system disorders) | 23
Neuropathy-motor (Nervous system disorders) | 26
Neuropathy-sensory (Nervous system disorders) | 66
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 25
Joint, pain (Musculoskeletal and connective tissue disorders) | 9
Muscle pain (Musculoskeletal and connective tissue disorders) | 7
Pain NOS (General disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less